CLINICAL TRIAL: NCT03419494
Title: Comparison of Remission Rate and Leukemic Stem Cell Changes Among Patients With Newly Diagnosed Adult ALL With Liposomal Doxorubicin and Daunorubicin-containing VDCLD Regimen.
Brief Title: Comparison of Liposomal Doxorubicin and Daunorubicin-containing VDCLD Regimen in the Treatment of Adult ALL Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013ALL-PLD
Record Dates: First submitted 2018-01-11; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Adult Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — 1-dodecylpyridoxal; liposomal doxorubicin; Daunorubicin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VDCLD regimen containing PLD: PLD 36mg/㎡.d d1、d15，ivdrip，1h，VCR 1.4mg/㎡.d d1，d8，d15，d22 iv，CTX 800mg/㎡.d d1 ivdrip，L-asp 6000u/㎡.d d19～28 ivdrip，Dex10mg.d d1～28 ivdrip
  Interventions: Drug: PLD
- VDCLD regimen containing DNR: DNR 45mg/㎡.d d1～3，ivdrip，1h，VCR 1.4mg/㎡.d d1，d8，d15，d22 iv，CTX 800mg/㎡.d d1 ivdrip，L-asp 6000u/㎡.d d19～28 ivdrip，Dex10mg.d d1～28 ivdrip
  Interventions: Drug: DNR

INTERVENTIONS:
Drug: PLD — PLD36mg/m2.d d1、d15，ivdrip，1h，VCR 1.4mg/m2.d d1，d8，d15，d22 iv，CTX 800mg/m2.d d1 ivdrip，L-asp 6000u/m2.d d19～28 ivdrip，Dex10mg.d d1～28 ivdrip
  Other Names: pegylated liposomal doxorubicin
  Groups: VDCLD regimen containing PLD
Drug: DNR — DNR 45mg/m2.d d1～3，ivdrip，1h，VCR 1.4mg/m2.d d1，d8，d15，d22 iv，CTX 800mg/m2.d d1 ivdrip，L-asp 6000u/m2.d d19～28 ivdrip，Dex10mg.d d1～28 ivdrip
  Other Names: Daunorubicin
  Groups: VDCLD regimen containing DNR

SUMMARY:
This trial is a multicenter prospective, open, non-intervention clinical study. 200 patients with newly diagnosed adult ALL who underwent induction remission with the VDCLD regimen containing PLD and DNR, respectively,were plan to enrolled in this study to evaluate the CR rate and the level of myeloid leukemia stem cells in the first course of chemotherapy with two regimens; and to evaluate the safety of the two induction chemotherapy regimens.

DETAILED DESCRIPTION:
Subjects will receive one of two treatment regimens:

Group A: intravenous drip of liposomal doxorubicin 36 mg/m2, d1、d15，1h； VCR 1.4mg/m2.d d1，d8，d15，d22 iv，CTX 800mg/m2.d d1 ivdrip，L-asp 6000u/m2.d d19～28 ivdrip，Dex10mg.d d1～28 ivdrip，once every 28days.

Group B: intravenous drip of DNR45mg/m2，d d1～3，1h；VCR 1.4mg/m2.d d1，d8，d15，d22 iv，CTX 800mg/m2.d d1 ivdrip，L-asp 6000u/m2.d d19～28 ivdrip，Dex10mg.d d1～28 ivdrip，once every 28days. The primary endpoint is complete remission after the first course treatment of induced remission chemotherapy, to evaluated the ratio of CR patients after the first course of chemotherapy with PLD and DNR VDCLD regimens.The secondary endpoint is to evaluate the changes of myeloid leukemia stem cells in patients before and after induction of VDCLD with PLD and DNR respectively.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female, age:14-60 years old; 2.ECOG score 0-2; 3.Subjects had confirmed ALL (WHO classification, primitive cells ≥ 20%); 4.Patients with newly diagnosed ALL who have not previously received chemotherapy (except for dexamethasone, prednisone, hydroxyurea).Blood transfusion, use of hematopoietic growth factors or vitamins are allowed. Some temporary measures such as leukocyte removal, dexamethasone, prednisone, hydroxyurea (0.5-3g daily, over 3 days) are allowed; 5.Flow cytometry was used to detect leukemic stem cells in bone marrow samples before treatment; 6.Informed consent (all studies must be signed patient informed consent).

Exclusion Criteria:

* 1.Mixed AL patients; 2.Active systemic infection; 3.Lactating women, fertile women with positive pregnancy tests for urine or pregnant women who are unwilling to adopt appropriate methods of contraception (such as the use of birth control pills, intrauterine devices, diaphragms, abstinence, condom use) during the study ; 4. Patients currently have a history of cardiac insufficiency (especially congestive heart failure) or previous history of congestive heart failure; 5. Patients with severe liver failure (≥5 times upper limit of normal transaminase, total bilirubin ≥3 mg/dL); 6. Patients had renal insufficiency with creatinine clearance <30 ml/min and creatinine clearance calculated as follows: Male: Ccr (ml / min) = (140-age) × body weight (kg) / [0.8136 × serum creatinine (μmol/L)] women: Ccr (ml/min) = (140-age) × body weight (kg) × 0.85 / [0.8136 × serum creatinine (μmol/L)]; 7. Patient is involved in other drugs experimental study within 30 days prior to the trial or within 90 days of the start of the trial; 8. Researchers think it is not suitable for enrolling.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This clinical trial will evaluate patients with primary adult ALL who meet the aboving inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-10-10 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
CR | From date of randomization until the date of first course of chemotherapy treatment completed, assessed up to 4 weeks.
  complete remission after the first course treatment of induced remission chemotherapy

SECONDARY OUTCOMES:
changes of myeloid leukemia stem cells | From date of randomization until the date of first course of chemotherapy treatment completed, assessed up to 4 weeks.
  to evaluate the changes of myeloid leukemia stem cells in patients before and after induction of VDCLD with PLD and DNR respectively.

CONTACTS AND LOCATIONS:
Overall Officials: zhigang yang, doctor, Principal Investigator — Affiliated Hospital of Guangdong Medical University
Locations (1):
- Affiliated Hospital of Guangdong Medical University, Guangdong, Guangdong, China